CLINICAL TRIAL: NCT01421992
Title: Phase 2/3 Study of Efficacy and Tolerability of Methylphenidate in the Treatment of Excessive Daytime Sleepiness in Myotonic Dystrophy Type 1
Brief Title: Methylphenidate in Myotonic Dystrophy Type 1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFM-12117; AFM-12117 (Other Grant/Funding Number: AFM-12117)
Record Dates: First submitted 2011-06-01; First posted 2011-08-23 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-06

CONDITIONS: Dystrophia Myotonica 1
Keywords: randomized; double-blind; crossover; methylphenidate; excessive daytime sleepiness
MeSH Terms: conditions — Myotonic Dystrophy; Disorders of Excessive Somnolence | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Methylphenidate versus baseline (Placebo Comparator)
  Interventions: Drug: Methylphenidate
- Arm 2: Placebo versus baseline (Placebo Comparator): One table placebo per day during 3 week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — One Tablet of methylphenidate, 20 mg per day during 3 weeks
  Other Names: Ritalin
  Arms: Arm 1: Methylphenidate versus baseline
Drug: Placebo — one tablet placebo per day during 3 weeks
  Arms: Arm 2: Placebo versus baseline

SUMMARY:
The purpose of this study is to determine whether methylphenidate is effective in the treatment of excessive daytime sleepiness due to myotonic dystrophy type 1 (DM1).

DETAILED DESCRIPTION:
Myotonic dystrophy type 1 (DM1) is a multisystemic disorder characterized by muscle weakness, myotonia, and the involvement of several systems. Hypersomnolence is one of the most frequently reported symptoms in patients with DM1 and often lead to handicap such as cessation of employment and withdrawal from social activities.The current investigation represents a prospective, double-blind, randomized, crossover, placebo-controlled study designed to evaluate the efficacy of methylphenidate for the treatment of excessive daytime sleepiness (EDS) in adults with DM1.

ELIGIBILITY:
Inclusion Criteria:

* adults
* Epworth score ≥ 10
* Diagnosis of myotonic dystrophy type 1

Exclusion Criteria:

* hypersensibility to methylphenidate
* Pregnancy
* Patients who receive drugs that interfere with methylphenidate
* Cognitive impairment
* Sleep apnea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline of excessive daytime sleepiness | 3 weeks after treatment

SECONDARY OUTCOMES:
Change from baseline of POMS, Rand36-Item Health survey and mean sleep latency | 3 weeks after treatment
  Mean sleep latency was measured using the behavioural Osler's test

CONTACTS AND LOCATIONS:
Overall Officials: Jack J Puymirat, MD, Principal Investigator — University Laval
Locations (1):
- Institute of Readaptation in Physical Deficiency, Québec, Quebec, Canada

REFERENCES:
- [Derived] Annane D, Laberge L, Gallais B, Chevret S. Psychostimulants for hypersomnia (excessive daytime sleepiness) in myotonic dystrophy. Cochrane Database Syst Rev. 2024 Nov 18;11(11):CD003218. doi: 10.1002/14651858.CD003218.pub3. PMID 39555632
- [Derived] Puymirat J, Bouchard JP, Mathieu J. Efficacy and tolerability of a 20-mg dose of methylphenidate for the treatment of daytime sleepiness in adult patients with myotonic dystrophy type 1: a 2-center, randomized, double-blind, placebo-controlled, 3-week crossover trial. Clin Ther. 2012 May;34(5):1103-11. doi: 10.1016/j.clinthera.2012.03.060. PMID 22578232